CLINICAL TRIAL: NCT00962702
Title: Exclusion of the Left Atrial Appendage With the LAAx, Inc., TigerPaw™ System During Elective, Non-Endoscopic Cardiac Surgery Procedures
Brief Title: Exclusion of the Left Atrial Appendage (LAA) With the LAAx, Inc. TigerPaw System
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LAAx, Inc. (Industry)
Responsible Party: William Wheeler, CEO LAAx,Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LAAx1DD20809
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Stroke
Keywords: Exclusion; Left Atrial Appendage; Surgical; Open chest
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exclusion of Left Atrial Appendage (Experimental): Exclusion of Left Atrial Appendage
  Interventions: Device: LAAx TigerPaw System

INTERVENTIONS:
Device: LAAx TigerPaw System — Exclusion of Left Atrial Appendage

SUMMARY:
The dual primary safety and effectiveness outcomes for the use of The TigerPaw System include the rate of device related adverse and serious adverse events and the extent of complete exclusion of the LAA with minimal residual cavity.

DETAILED DESCRIPTION:
The primary safety outcome is the rate of device related adverse and serious adverse events assessed peri-operatively, and at 30 and 90 days post procedure. The primary effectiveness outcome is the percentage of patients with complete exclusion of the left atrial appendage assessed peri-operatively (visually), and at 90 days post procedure via transesophageal echocardiography (TEE).

Transesophageal echocardiography will be performed intra-operatively and again at 90 days post procedure. Intra-operative and follow-up TEE examinations will be read centrally at a core laboratory. Any Doppler flow across the Fastener into the excluded portion of the appendage will also be considered a failure of exclusion. The presence or absence of LAA and/or LA thrombus will be evaluated. Patients will also be evaluated for other potential sources of embolism, including aortic atheroma, patent foramen ovale, or other intracardiac shunts.

Data collection will be completed at baseline, at the time of open cardiac surgery procedure and throughout the perioperative hospitalization. Patients will be evaluated at 30 days post surgery and at 90 days post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years of age
2. Stroke Risk (CHADS score > or = 2, CHADS scoring: CHF = 1 pt, Hypertension (or treated hypertension) = 1 pt, Age > 75 = 1 pt, Diabetes = 1 pt, Prior stroke or TIA = 2 pts)
3. Subject scheduled to undergo elective non-endoscopic cardiac surgical procedure(s) including cardiac surgery for one or more of the following:

   * mitral valve repair or replacement
   * aortic valve repair or replacement
   * tricuspid valve repair or replacement
   * coronary artery bypass procedures
   * concomitant surgical (ablation or cut and sew) Maze procedure
4. Ejection fraction > 30%
5. Absence of thrombus in LAA
6. During open procedure, LAA anatomy is determined to be suitable for closure
7. life expectancy of > 1 year
8. patient willingness to cooperate with follow-up tests
9. Informed Consent

Exclusion Criteria:

1. Previous cardiac surgery
2. Contraindication to Transesophageal Echocardiography (TEE)
3. Thrombus in the LAA/LA
4. NYHA Class IV heart failure symptoms
5. Need for emergent cardiac surgery (e.g., cardiogenic shock)
6. Creatinine > 200 umol/L
7. Current diagnosis of active systemic infection
8. Renal failure requiring dialysis or hepatic failure
9. A known drug and/or alcohol addiction
10. mental impairment or other conditions which may not allow the subject to understand the nature, significance and scope of the study and to cooperate with follow-up requirements
11. Preoperative need for an intra-aortic balloon pump or intravenous inotropes
12. Treatment with thoracic radiation
13. Concurrent chemotherapy
14. Long term treatment with steroids not including intermittent use of inhaled steroids for respiratory diseases
15. Known connective tissue disorders
16. Coagulation disorders
17. Any active medical condition that would preclude the patient from completing the study or would result in an unreasonable risk
18. Active participation in another clinical trial.
19. Intraoperative:

    * LAA is not appropriate for exclusion based upon intraoperative evaluations
    * Presence of thrombus in LAA or LA; or
    * Any other findings by surgeon/investigator that would preclude use of device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-12 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
The dual primary safety and effectiveness outcomes include the rate of device related adverse and serious adverse events and the extent of complete exclusion of the LAA with minimal residual cavity. | Patients will be evaluated at 30 days post surgery and at 90 days post surgery.

SECONDARY OUTCOMES:
The extent of complete exclusion of the LAA with minimal residual cavity. | 30 days post surgery and at 90 days post

CONTACTS AND LOCATIONS:
Overall Officials: Mark Slaughter, MD, Principal Investigator — University of Louisville
Locations (1):
- Clarian Health / Methodist Hospital, Indianapolis, Indiana, United States